CLINICAL TRIAL: NCT06712108
Title: PROspective Multicenter Observational Study of Double Unit Umbilical Cord Lood Transplantation in Korean Adult Patients With Hematologic Diseases.
Brief Title: Double Unit Cord Blood Transplant in Hematologic Malignancies.
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong-Yeop Shin, Associate Professor, Seoul National University Hospital
Other Study IDs: PRODUCT-K
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adult Double Unit Cord Blood Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — cord blood bone marrow and peripheral blood samples at follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with hematologic disease who will receive double unit cord blood tranplant
  Interventions: Procedure: tranplant

INTERVENTIONS:
Procedure: tranplant — double unit cord blood transplnat

SUMMARY:
The efficacy and safety of non-myeloablative and myeloablative preconditioning followed by dual-unit umbilical cord blood transplantation from unrelated donors in adult patients with malignant hematologic diseases eligible for allogeneic hematopoietic stem cell transplantation are evaluated through prospective observation and analysis of actual clinical data collection

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 and older
* Patients scheduled for umbilical cord blood transplantation as a primary allogeneic hematopoietic stem cell transplantation for the treatment of the following hematologic diseases:

Acute leukemia (myeloid/lymphoid/mixed lineage) / Myelodysplastic syndromes / Chronic leukemia (myeloid/lymphoid/monocytic) and myeloproliferative neoplasms / Malignant lymphomas, multiple myeloma / Other malignant hematologic malignancies / bone marrow failure diseases, including aplastic anemia

- If all contents of the consent form are understood and consented to in writing.

Exclusion Criteria:

* Patients with a history of allogeneic hematopoietic stem cell transplantation or those undergoing transplantation for the treatment of engraftment failure (secondary allogeneic hematopoietic stem cell transplantation is an exclusion criterion; however, patients eligible for registration include those undergoing their first allogeneic stem cell transplantation following an autologous stem cell transplantation).
* Patients with severe, uncontrolled infections or severe cardiopulmonary dysfunction, as judged by the investigator.
* Patients with an ECOG Performance Status (PS) greater than 3 or those receiving mechanical ventilation in the intensive care unit.
* Patients who do not consent to participate in the study or those deemed unsuitable for sincere participation by the attending physician.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with malignant hematologic diseases who are eligible for allogeneic hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years

SECONDARY OUTCOMES:
engraftment | 30 days
  Frequency of engraftment
GVHD | 2 years
  acute and chronic GVHD
PFS | 2 years
  Progression-free survival
TRM | 3 months
  Treatment related mortality
Relapse | 2 years
  Relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Yeop Shin, MD, PhD., Principal Investigator — Seoul National University Hospital; Sung-Soo Yoon, MD, PhD., Study Director — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Jeonbuk National University Hopital, Jeonju, Jeonlabuk-do
  - Keimyung Unversity Dongsan Hospital, Daegu
  - Dong-A University Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No